CLINICAL TRIAL: NCT06972420
Title: Improving the Quality of Anesthesia Induction by Reducing Preoperative Anxiety in the Operating Room
Acronym: QUALIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A02469-38
Record Dates: First submitted 2025-04-15; First posted 2025-05-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Anxiety at Induction of Pediatric Anesthesia
Keywords: Anxiety at induction; Preoperative anxiety

STUDY DESIGN:
Intervention Model Description: The study is a monocentric, pilot, exploratory, open-label, prospective quasi-experimental "before/after" study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 2: Standard preoperative care before anesthesia induction (No Intervention): Part 2: Children aged between 5 and 12 years scheduled for surgery requiring hospitalization, recieving standard preoperative care prior to anesthesia induction. Anxiety levels will be measured at the time of induction in the operating room.
- Parti 1: Preoperative care combined with a hypnosis session (Experimental): Part 1: Children aged between 5 and 12 scheduled for surgery requiring hospitalization, recieving a 20 min hypnosis session within two weeks prior to anesthesia induction in addition to standard preoperative care. Anxiety levels will be measured at the time of induction in the operating room.
  Interventions: Behavioral: Hypnosis session

INTERVENTIONS:
Behavioral: Hypnosis session — Within the two weeks prior to surgery, in addition to the standard preoperative care currently in place, the patient will receive a 30-minute visit from a nurse anesthetist trained in hypnosis. This is an added procedure complementing the anesthesia consultation. The visit is divided into two parts: 10 minutes to review and clarify the explanations given by the anesthesiologist and surgeon, and 20 minutes of a formal hypnosis session. A personalized liaison form will be completed to facilitate communication between the consultation and the operating room.
  Arms: Parti 1: Preoperative care combined with a hypnosis session

SUMMARY:
Preoperative anxiety refers to a range of physical and/or psychological manifestations, which can have a significant impact on medical outcomes and the experience of the child and their parents. This study aims to evaluate the impact of preoperative preparation combined with a hypnosis session conducted by nurse anesthetists (IADE) trained in working with children and their families. The goal is to improve the child's experience and reduce perioperative anxiety and stress.

It is divided into two phases:

* First phase, called "Before": Standard preoperative care is provided according to the existing protocol in the department. Anxiety levels will be measured at the time of induction in the operating room.
* Second phase, called "After": In the two weeks prior to surgery, in addition to the standard preoperative care currently in place, the patient will receive a 30-minute visit from a nurse anesthetist trained in hypnosis. This is an added procedure complementing the anesthesia consultation. The visit is divided into two parts: 10 minutes to review and clarify the explanations given by the anesthesiologist and surgeon, and 20 minutes of a formal hypnosis session. A personalized liaison form will be completed to facilitate communication between the consultation and the operating room. Anxiety levels will again be measured at the time of induction.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 5 and 12 years, i.e., able to engage in verbal communication;
* Scheduled for surgery requiring hospitalization at least one day prior to the procedure, including but not limited to gastrointestinal or urological surgery, ENT procedures, plastic interventions, and orthopedic surgery (e.g., scoliosis correction);
* Provision of written informed consent by the parents or legal guardians (or by the sole parent/legal guardian, where applicable);
* Parental agreement to participate in the study by completing the required questionnaires;Affiliation with or entitlement to a national social security scheme

Exclusion Criteria:

* Patients with cognitive developmental disorders;
* Patients requiring regular general anesthesia as part of ongoing medical management;
* Patients undergoing emergency surgery;
* Patients with a known psychiatric disorder;
* Patients diagnosed with an autism spectrum disorder (ASD).

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2026-10-02 (Estimated)

PRIMARY OUTCOMES:
Children's perioperative anxiety levels at the time of anesthetic induction as assessed by the mYPAS | Day 1 ( Anesthesia induction and surgery)
  Mesure of the Modified Yale Preoperative Anxiety Scale by anesthetics or surgical nurse. The total score ranges from 23 to 100: children are considered moderately anxious for a score above 24, and highly anxious for a score above 30.

SECONDARY OUTCOMES:
Children's compliance during induction as assessed by the Induction Compliance Checklist | Day 1 (Anesthesia induction)
  Induction compliance check list at the time of anesthetic induction
Time spent in the PACU | Day 1 ( From arrival in the PACU until return to the hospital room)
  Duration in minutes between arrival in the PACU and return to the hospital room
Postoperative delirium as assessed by the PAED Scale | Day 1 (After surgery)
  Assessed in the PACU using the PAED scale (Pediatric Anesthesia Emergence Delirium).
Postoperative pain as assessed by the VAS scale | Day 1 (After surgery)
  Evaluated in the recovery room using the Visual Analogue Scale (VAS). Total scole ranging from 0 to 10 where a higher scores mean worse pain.
Postoperative pain as assessed by the FLACC scale. | Day 1 (After surgery)
  Evaluated in the recovery room using the Face Legs Activity Cry Consolability (FLACC) scale. Total scole ranging from 0 to 10 where a higher scores mean worse pain.
Postoperative pain as assessed by the PPMP scale | Day 2 and 5 after sugery
  Assessed by parents on postoperative days 2 and 5 using the Parents' Postoperative Pain Measure (PPPM), either during hospitalization or via telephone follow-up. The score ranges from 0 to 15, where a higher scire mean worse pain
Behavioral assessment | Day 1, 2 and 5 after sugery
  The child's postoperative behavior will be assessed on postoperative days 2, 5, and 14 using the PHBQ (Post-Hospitalization Behavior Questionnaire), either in the hospital or via a phone call.
Parental satisfaction | At the day of patiet sicharge or Day 14 postoperatevly
  Assessed via a dedicated questionnaire, either in the hospital or through a phone call

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No